CLINICAL TRIAL: NCT06170060
Title: Preventing and Treating Reflux With Cruroplasty and Omentopexy After Laparoscopic Sleeve Gastrectomy
Brief Title: Treatment of Reflux With Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yusuf Emre ALTUNDAL (Other)
Responsible Party: Sponsor-Investigator, Yusuf Emre ALTUNDAL, Assistant Professor, Istanbul Aydın University
Organization: Istanbul Aydın University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAU-YUSUFEMREALTUNDAL-001
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Reflux Disease, Gastro-Esophageal; Hiatal Hernia; Reflux Esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal; Esophagitis, Peptic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic Sleeve Gastrectomy (Experimental)
  Interventions: Other: Laparoscopic Sleeve Gastrectomy

INTERVENTIONS:
Other: Laparoscopic Sleeve Gastrectomy — Laparoscopic sleeve gastrectomy (LSG) is a surgical procedure widely used in the treatment of obesity. It's a bariatric procedure, meaning its primary aim is to induce weight loss, and it has gained popularity due to its effectiveness and relatively low complication rates compared to other bariatric surgeries.

SUMMARY:
In 2008, the World Health Organization (WHO) report found that 0.5-1.5 billion people aged 20 years and above suffer from overweight (body mass index (BMI) ≥ 25) and obesity (BMI ≥ 30 kg / m2) stated.

WHO estimates that the number of overweight and obese people will reach 2.3 and 0.7 billion, respectively, by 2045.

Bariatric surgery has been developed in response to the number of obese patients living in the world and the complications caused by obesity. The most common type of bariatric surgery against obesity is Laparoscopic Sleeve Gastrectomy (LSG).

As after any surgical operation, complications may occur after Laparoscopic Sleeve Gastrectomy. Additional operations may be required to correct complications such as bleeding, anastomotic leak, gastric volvulus, infection, dyspepsia, hiatal hernia, bile and/or acid reflux.

The incidence of gastroesophageal reflux disease (GERD) is significantly increased in obese patients compared to the incidence in normal individuals. Various studies have shown that obesity causes delayed gastric emptying due to increased abdominal pressure, esophageal motility disorders, especially hypotensive lower esophageal sphincter pressure (<10 mm Hg), finally the development of hiatal hernia (HH), whose prevalence in the obese population is significantly higher than in non-obese patients.

Various surgical methods have been presented to prevent postoperative de-novo Gastroesophageal Reflux and de-novo Hiatal Hernia that occur after LSG. Curorrhaphy is one of these techniques that is accepted to prevent the formation or exacerbation of postoperative GERD and Hiatal Hernia.

In this surgical technique, after the diaphragmatic crura are completely exposed at the level of the lower esophageal sphincter (LES), the hiatal hernia, if present, is reduced into the abdomen. Afterwards, Z surgical sutures are applied to the diaphragmatic crura to make the diaphragmatic esophageal ring narrow enough. In this way, it is aimed to strengthen the diaphragmatic crus. Findings following cruroplasty for GERD prevention are varied. Although some authors state that the technique does not provide an advantage in preventing postoperative GERD, some studies have shown cruroplasty to be effective.

In this study, investigators aimed to show that the technique of simultaneous cruroplasty and single suture omentopexy with LSG is a treatment for GERD and HH, which are very common in obese patients, and a preventive technique for de-novo GERD seen after LSG.

ELIGIBILITY:
Inclusion Criteria:

* Obesity,

Exclusion Criteria:

* Eating disorder or mental disorder
* Misunderstanding of the protocol
* Psychiatric contraindication
* Patient participating in another interventional clinical research protocol involving a drug or medical device
* Pregnant, breastfeeding

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
The Gastroesophageal Reflux Disease Health-Related Quality of Life Survey | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Küçükçekmece, Istanbul, Turkey (Türkiye)